CLINICAL TRIAL: NCT06089057
Title: Activation for Self-Care Needs in Older Adults With Chronic Kidney Disease: ACTIVE SENIORS With CKD
Brief Title: Pro-social Power Training Activity for Aging and Well-being With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NEPH-007-23S; 1IK2CX002595-01A2 (NIH)
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Lower Extremity Muscle Strength
Keywords: mobility
MeSH Terms: interventions — Aging; Health

STUDY DESIGN:
Intervention Model Description: Veterans will be randomized to either the intervention to an attention control. Randomization will be performed by the biostatistician. Veterans will be randomized to the intervention group (or to the attention control) using a block randomization scheme with randomly selected block sizes of 2, 4, and 6. Participants in the attention control will receive educational resources regarding the benefits of physical activity prior to intervention start (A brief document related to the importance of physical activity in kidney disease and handouts from the Center for Disease Control's recommendations for physical activity for older adults). Participants in the attention control may also receive a weekly phone call on general health.
Who Masked: Outcomes Assessor
Masking Description: All research assistants and biostatistics personnel will be masked to each participant's assignment. Participants and study staff are unaware of group allocation at the time of recruitment and baseline assessments because randomization is performed after participants have completed baseline assessments. However, there is no blinding to group allocation after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Power training and monitored physical activity (Experimental): This is a 16-week power-training and physical activity-focused intervention that contains in-center and at-home components and motivational coaching. Participants will meet 2-3 times per week for the in-center power training. Participants will also be asked to wear accelerometers at home in order for their physical activity frequency to be measured.
  Interventions: Behavioral: Pro-social Power training Activity for Aging and Well-being with Chronic Kidney Disease
- Attention control (Active Comparator): This will be the attention control arm that will involve receipt of a physical activity education booklet, use of an accelerometer, and weekly check-in calls. No power training or motivational coaching will be delivered.
  Interventions: Behavioral: Attention Control for Pro-social Power training Activity for Aging and Well-being with Chronic Kidney Disease

INTERVENTIONS:
Behavioral: Pro-social Power training Activity for Aging and Well-being with Chronic Kidney Disease — This is a 16-week power-training and physical activity-focused intervention that contains group in-center and individual at-home components and motivational coaching. Participants will meet 2-3 times per week for the in-center power training. Participants will also be asked to wear accelerometers at home in order for their physical activity frequency to be measured.
  Other Names: PACT to AGE WELL with CKD
  Arms: Power training and monitored physical activity
Behavioral: Attention Control for Pro-social Power training Activity for Aging and Well-being with Chronic Kidney Disease — This will be the attention control arm that will involve receipt of a physical activity education booklet, use of an accelerometer, and weekly check-in calls. No power training or motivational coaching will be delivered.
  Other Names: Attention Control for PACT to AGE WELL with CKD
  Arms: Attention control

SUMMARY:
This is a pilot trial of a 16-week physical activity and power training program among 30 Veterans/arm with advanced chronic kidney disease. The trial aims to test whether the program is tolerable to Veterans.

DETAILED DESCRIPTION:
This will be a randomized controlled pilot trial of a 16-week physical activity and power training intervention trial among 30 pre-frail Veterans with Stage 3B-5 chronic kidney disease. The intervention will contain in-center and at-home components. It will lay the foundation for a large-scale future randomized controlled efficacy trial aimed to reduce frailty risk among Veterans with advanced chronic kidney disease. 30 other Veterans will be part of an attention control.

The outcomes of this pilot trial are feasibility, acceptability, and fidelity. Each of these outcomes will be measured using quantitative surveys and data review as well as qualitative assessments among Veterans at trial close. As this is a pilot feasibility trial, it is intentionally not powered to detect whether the intervention has a significant effect on physical activity frequency, muscle strength, or physical frailty.

ELIGIBILITY:
Inclusion Criteria:

* Participant's nephrologist and/or primary care physician agree that participant may enroll in trial
* Participants classified as pre-frail per Fried Frailty phenotype due to slowness (time taken to walk 15 feet is greater than 6 seconds) in Aim 1, OR who report 'YES' to any of the following:

  * "For health or physical reasons, do you have difficulty in walking a mile (5-6 blocks)?", OR
  * "If no, have you changed the way you walk half a mile (5-6 blocks) because of underlying health problems?", OR
  * "For health or physical reasons, do you have difficulty in climbing 1 flight of stairs (10 steps)?", OR
  * "If no, have you changed the way you climb 1 flight of stairs (10 steps) because of health problems?"

Exclusion Criteria:

* Myocardial infarction or unstable angina within the prior six months based on electronic medical record review or self-report
* Uncontrolled cardiac arrythmia within the prior six months based on electronic medical record review or self-report
* Systolic blood pressure > 180 mm Hg and/or diastolic blood pressure > 110 mm Hg on more than one occasion within prior six months based on electronic medical record review or self-report
* Cerebrovascular event and/or transient ischemic attack within prior six months based on electronic medical record review or self-report
* Abnormal cardiac stress test within the past year based on electronic medical record review or self-report
* Hemoglobin of 10 g/dL or less based on electronic medical record review or self-report
* Class IV heart failure based on electronic medical record review or self-report
* Dyspnea and/or chest pain at rest
* Dependence on wheelchair for mobility
* Permanent residence in nursing home or other long-term care facility
* Terminal illness or other hospice-qualifying medical condition
* Planned move away from middle Tennessee within the next year
* Planned major surgery in the next six months
* Blindness
* Concurrent enrollment in physical therapy or structured exercise program
* Anticipated dialysis or kidney transplant in upcoming three months
* Non-English speaking
* Severe cognitive impairment based on electronic medical record review or self-report

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility, as measured by the questionnaire, the Feasibility of Intervention Measure | 4 months
  This will be a brief questionnaire known as the Feasibility of Intervention Measure, that asks participants whether the intervention seems doable to them. There are four questions, and participants are asked to rate intervention feasibility from a scale of 1 (Strongly Disagree) to 5 (Strongly Agree). Scores range from 1-5 and are calculated as the mean of all scores. Higher scores indicate greater perceived feasibility. This will not be aggregated with any other measure.
Feasibility, as measured by a numerical percentage of all participants who consented out of those eligible | 4 months
  This will be a numeric percentage of participants who consent for the pilot trial out of all eligible participants in Aim 1. This will not be aggregated with any other measure.
Feasibility, as measured by a qualitative description of participants' reasons for declining | 4 months
  This will be a qualitative description of potential participants' reasons for declining, if applicable. This will not be aggregated with any other measure.

OTHER OUTCOMES:
Acceptability, as measured by the questionnaire, the Acceptability of Intervention Measure | 4 months
  This will be a brief questionnaire known as the Acceptability of Intervention Measure, that asks participants whether the intervention seems acceptable and/or enjoyable to them. There are four questions, and participants are asked to rate intervention acceptability from a scale of 1 (Strongly Disagree) to 5 (Strongly Agree). Scores range from 1-5 and are calculated as the mean of all scores. Higher scores indicate greater perceived acceptability. This will not be aggregated with any other measure.
Acceptability, as measured by participants' qualitative descriptions of reasons for intervention enjoyability, if applicable | 4 months
  This will be a qualitative description of participants' reasons they found the intervention enjoyable to participate in, if applicable. This will not be aggregated with any other measure.
Fidelity, as measured by the percentage of sessions participants attended out of all possible sessions | 4 months
  This will be a percentage, measured by the number of sessions a participant attended out of all possible sessions that could have have been attended. This will not be aggregated with any other measure.
Fidelity, as measured by accelerometer step count during prior week | 5 months, 6 months, and 7 months
  This will be the step count during the prior week recorded on an accelerometer worn by each participant. This will be measured at each of the following time points: one, two, and three months after intervention close. That is to say, this will be measured at 5 months, 6 months, and 7 months after intervention start. This will not be aggregated with any other measure.
Fidelity, as measured by the questionnaire, the Physical Activity Scale for the Elderly | 5 months, 6 months, and 7 months
  This will be measured using the questionnaire, the Physical Activity Scale for the Elderly, a ten-item questionnaire that inquires about the frequency, duration, and intensity of physical activity during the prior week. Scores range from 0-793, with higher scores indicating completion of more frequent and/or intense physical activity. This will be measured at each of the following time points: one, two, and three months after intervention close. That is to say, this will be measured at 5 months, 6 months, and 7 months after intervention start. This will not be aggregated with any other measure.
Fidelity, as measured by participants' descriptions of reasons for adherence vs. nonadherence | 7 months
  This will be a qualitative description of participants' reasons for adhering to the intervention or not, as applicable. This will not be aggregated with any other measure.
Adverse events, as measured by the the number of participants who report adverse events from the Common Terminology Criteria for Adverse Events, v5.0 | 7 months
  This will be the total number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 5.0. This will not be aggregated with any other measure.
Adverse events, as measured by the type of adverse events reported on the Common Terminology Criteria for Adverse Events, v5.0 | 7 months
  This will be the type of adverse events as reported by participants from the Common Terminology Criteria for Adverse Events version 5.0. This will not be aggregated with any other measure.

CONTACTS AND LOCATIONS:
Overall Officials: Devika Nair, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (1):
- Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No